CLINICAL TRIAL: NCT04217187
Title: The Effect of Electrical Stimulation Post Botulinum Toxin Injections on Functional Use of the Hemiparetic Upper Extremity
Brief Title: Electrical Stimulation After Botulinum Toxin Injections to the Upper Extremity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas Woman's University (Other)
Collaborators: TIRR Memorial Hermann (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-FY2020-43
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Stroke
Keywords: Botulinum Toxins; Spasticity; Upper Extremity; Electrical Stimulation
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electrical Stimulation Group (Experimental): This arm will receive neuromuscular electrical stimulation to the antagonist muscles of the upper extremity.
  Interventions: Device: Neuromuscular Electrical Stimulation
- Sham Stimulation Group (Sham Comparator): This arm will receive sensory stimulation without muscle contraction to the antagonist muscles of the upper extremity.
  Interventions: Device: Sham Electrical Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Upper extremity neuromuscular electrical stimulation
  Arms: Electrical Stimulation Group
Device: Sham Electrical Stimulation — Sensory only upper extremity electrical stimulation
  Arms: Sham Stimulation Group

SUMMARY:
The purpose of this study is to investigate the effectiveness of using electrical stimulation to improve upper extremity function in stroke survivors who receive botulinum toxin injections for spasticity. We hypothesize that individuals who receive the electrical stimulation could demonstrate improved benefit of the botulinum toxin injections and improved functional use of their weaker upper extremity.

DETAILED DESCRIPTION:
This is a pragmatic investigation that will utilize a two group comparison to compare electrical stimulation to a sham stimulation in individuals who are scheduled to receive botulinum toxin injections to their upper extremity for spasticity management. The electrical stimulation will be to the antagonist muscles of the injected muscles of the upper extremity and will be administered for 4 weeks post injections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke, within first 6 months post stroke, have not previously received botulinum toxin injections for upper extremity spasticity, hemiplegic upper extremtity, able to communicate in English.

Exclusion Criteria:

* contraindication for electrical stimulation (presence of implanted cardiac or other medical device, open wound on the wrist or hand, malignancy), fixed contracture of the elbow, wrist or hand, inability to follow simple directions, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-01-13 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Chedoke-McMaster Stroke Assessment Measure- Arm and Hand Recovery Stage | Baseline, 1 month and 6 months after injections
  Impairment level assessment to measure changes in active motor control and isolated movement in the upper extremity. The arm and the hand receive a separate score. The score ranges from 1 to 7. A higher score indicates better arm function.

SECONDARY OUTCOMES:
Action Research Arm Test | Baseline, 1 month and 6 months
  Standardized measure of upper extremity function. The total score ranges from 0-57. A higher score indicates better arm function.
Box and Block Test | Baseline, 1 month and 6 months after injections
  Standardized measure of upper extremity function. The score is the number of blocks transported within one minute. A higher score indicates better arm function.
Motor Activity Log | Baseline, 1 month and 6 months after injections
  Structured interview to measure perceived function of the upper extremity during daily tasks. There is a separate score for the amount of use and how well measures. Each scale ranges from 0-5 and a higher score indicates better arm function.
Modified Ashworth Scale for the Upper Extremity | Baseline, 1 month and 6 months
  Measure of spasticity. Each muscle group (i.e. elbow flexors) is scored from 0-4 with a 0 indicating no increase in muscle tone and a 4 indicating the affected part is rigid. A decrease in score indicates a decrease in spasticity.
Numeric Pain Rating Scale | Baseline, 1 month and 6 months
  Self report of current, best and worst pain of upper extremity in the past 24 hours. Scale ranges from 0-10 with a 0 indicating no pain and a 10 indicating severe pain. A decrease in score indicates less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine C Hay, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- TIRR Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Bejot Y, Daubail B, Giroud M. Epidemiology of stroke and transient ischemic attacks: Current knowledge and perspectives. Rev Neurol (Paris). 2016 Jan;172(1):59-68. doi: 10.1016/j.neurol.2015.07.013. Epub 2015 Dec 21. PMID 26718592
- [Background] Parker VM, Wade DT, Langton Hewer R. Loss of arm function after stroke: measurement, frequency, and recovery. Int Rehabil Med. 1986;8(2):69-73. doi: 10.3109/03790798609166178. PMID 3804600
- [Background] Gracies JM. Pathophysiology of spastic paresis. I: Paresis and soft tissue changes. Muscle Nerve. 2005 May;31(5):535-51. doi: 10.1002/mus.20284. PMID 15714510
- [Background] Hebert D, Lindsay MP, McIntyre A, Kirton A, Rumney PG, Bagg S, Bayley M, Dowlatshahi D, Dukelow S, Garnhum M, Glasser E, Halabi ML, Kang E, MacKay-Lyons M, Martino R, Rochette A, Rowe S, Salbach N, Semenko B, Stack B, Swinton L, Weber V, Mayer M, Verrilli S, DeVeber G, Andersen J, Barlow K, Cassidy C, Dilenge ME, Fehlings D, Hung R, Iruthayarajah J, Lenz L, Majnemer A, Purtzki J, Rafay M, Sonnenberg LK, Townley A, Janzen S, Foley N, Teasell R. Canadian stroke best practice recommendations: Stroke rehabilitation practice guidelines, update 2015. Int J Stroke. 2016 Jun;11(4):459-84. doi: 10.1177/1747493016643553. Epub 2016 Apr 14. PMID 27079654
- [Background] Richardson D, Sheean G, Werring D, Desai M, Edwards S, Greenwood R, Thompson A. Evaluating the role of botulinum toxin in the management of focal hypertonia in adults. J Neurol Neurosurg Psychiatry. 2000 Oct;69(4):499-506. doi: 10.1136/jnnp.69.4.499. PMID 10990511
- [Background] Foley N, Pereira S, Salter K, Fernandez MM, Speechley M, Sequeira K, Miller T, Teasell R. Treatment with botulinum toxin improves upper-extremity function post stroke: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2013 May;94(5):977-89. doi: 10.1016/j.apmr.2012.12.006. Epub 2012 Dec 19. PMID 23262381
- [Background] Hesse S, Reiter F, Konrad M, Jahnke MT. Botulinum toxin type A and short-term electrical stimulation in the treatment of upper limb flexor spasticity after stroke: a randomized, double-blind, placebo-controlled trial. Clin Rehabil. 1998 Oct;12(5):381-8. doi: 10.1191/026921598668275996. PMID 9796928
- [Background] Hesse S, Jahnke MT, Luecke D, Mauritz KH. Short-term electrical stimulation enhances the effectiveness of Botulinum toxin in the treatment of lower limb spasticity in hemiparetic patients. Neurosci Lett. 1995 Dec 1;201(1):37-40. doi: 10.1016/0304-3940(94)12124-9. PMID 8830307
- [Background] Picelli A, Smania N, Storti I, Munari D, Fontana C, Fiaschi A, Santilli V, Tamburin S. Immediate versus delayed electrical stimulation boosts botulinum toxin effect: A pilot study. Mov Disord. 2011 Aug 1;26(9):1784-5. doi: 10.1002/mds.23678. Epub 2011 Apr 29. No abstract available. PMID 21538521
- [Background] Lee JM, Gracies JM, Park SB, Lee KH, Lee JY, Shin JH. Botulinum Toxin Injections and Electrical Stimulation for Spastic Paresis Improve Active Hand Function Following Stroke. Toxins (Basel). 2018 Oct 25;10(11):426. doi: 10.3390/toxins10110426. PMID 30366407
- [Background] Sheean GL. Botulinum treatment of spasticity: why is it so difficult to show a functional benefit? Curr Opin Neurol. 2001 Dec;14(6):771-6. doi: 10.1097/00019052-200112000-00015. PMID 11723387